CLINICAL TRIAL: NCT06946940
Title: Biosignature of the Response to Treatment With Cannabis Oil in Individuals With Fibromyalgia
Acronym: CAN-RCT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Collaborators: American Fibromyalgia Syndrome Association (Other)
Responsible Party: Principal Investigator, Amir Minerbi MD, Director, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0576-22
Record Dates: First submitted 2025-04-01; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Microbiome; Cannabis; Chronic Pain
MeSH Terms: conditions — Fibromyalgia; Marijuana Abuse; Chronic Pain | interventions — nabiximols

STUDY DESIGN:
Intervention Model Description: A Double-Blinded, Randomized Placebo-Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Comparator: Cannabis Oil (5% THC/5% CBD) (Active Comparator): Participants in this arm will receive cannabis oil containing a balanced formulation of 5% THC and 5% CBD. The intervention will span three months, including a six-week titration period to optimize dosing, followed by a maintenance phase. Doses will be self-administered sublingually and adjusted based on individual tolerance and efficacy. Comprehensive assessments will monitor clinical outcomes, gut microbiome composition, and circulating metabolomics to explore correlations with treatment response and safety.
  This arm will comprise 120 patients.
  Interventions: Drug: Cannabis Oil (5% THC/5% CBD)
- Sham Comparator: Placebo Oil (Sham Comparator): Participants in this arm will receive placebo oil, which is visually and chemically matched to the active cannabis oil but contains no active cannabinoids (THC or CBD). Like the active arm, participants will undergo a three-month intervention, including a six-week titration period and maintenance phase. Outcomes, including clinical measures and biological analyses, will be used as a control to evaluate the therapeutic effects of the cannabis oil.
  This arm will comprise 30 patients.
  Interventions: Drug: Sham Cannabis Oil

INTERVENTIONS:
Drug: Cannabis Oil (5% THC/5% CBD) — Cannabis oil containing a balanced formulation of 5% tetrahydrocannabinol (THC) and 5% cannabidiol (CBD). Administered sublingually over a three-month period, starting with a six-week titration phase to optimize dosing, followed by maintenance.
  Arms: Active Comparator: Cannabis Oil (5% THC/5% CBD)
Drug: Sham Cannabis Oil — Placebo oil visually and chemically matched to the active cannabis oil but devoid of active cannabinoids (THC/CBD). Administered sublingually over three months, mirroring the active arm's titration and maintenance schedule.
  Arms: Sham Comparator: Placebo Oil

SUMMARY:
Fibromyalgia is a chronic condition that causes widespread pain, fatigue, and other symptoms, significantly affecting quality of life. Unfortunately, there are few effective treatments available. Recently, medical cannabis has gained attention as a potential treatment, leading many countries to approve its use for fibromyalgia. However, its success is limited-only about 25% of patients experience meaningful pain relief, and side effects like dizziness or fatigue are common. Not everyone responds to medical cannabis the same way, and researchers think this variability may partly be explained by differences in the gut microbiome-the community of bacteria and other microorganisms living in our digestive system. These microbes are known to influence various aspects of health, including pain and how the body processes medications. Our research focuses on understanding the link between the gut microbiome and fibromyalgia. We propose a study where 150 fibromyalgia patients will be treated with either cannabis oil or a placebo in a double-blind trial. By analyzing their symptoms and gut microbiome, we hope to identify patterns that could predict who will benefit most from cannabis treatment. If successful, this research could lead to more personalized and effective treatment options for fibromyalgia.

DETAILED DESCRIPTION:
This study aims to explore the potential association between the composition of the gut microbiome and the individual response to cannabis oil in individuals with fibromyalgia. We propose a double-blinded randomized controlled trial, where 150 patients with fibromyalgia will be treated with either a careful titration of cannabis oil (5% THC, 5% CBD) or placebo with an allocation ratio of 4:1. Patient reported outcomes, quantitative sensory testing and gut microbiome and metabolome composition will be evaluated at baseline and during treatment. Subjective and objective clinical outcomes will be compared to baseline and end-of-study gut microbiome composition and metabolomic profile.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women aged 30 years and over.
* Diagnosis of fibromyalgia confirmed according to the 2016 diagnostic criteria by a pain specialist, with relevant symptoms lasting 12 months or more.
* An average reported pain ≥ 6 during the preceding week.
* Eligible for cannabis at the discretion of the treating physician.
* Has remained symptomatic despite receiving standard care for fibromyalgia including analgesics, anti-depressants (tricyclic and SNRI) and anti-epileptic agents.

Exclusion Criteria:

* Patients who have used cannabis during the preceding month.
* Any significant comorbid condition at the discretion of the PI (e.g. inflammatory arthritis, inflammatory bowel disease, cancer).
* Personal or family history of psychotic disorders.
* Current or past anxiety disorder.
* Any uncontrolled psychiatric pathology.
* Current or history of substance addiction or abuse.
* Diagnosed dementia or cognitive impairment.
* Personal history of cardiovascular disease.
* Pregnancy, lactation or intention to conceive.
* Known allergy to any of the cannabis oil ingredients.
* Patients with a history of seizure disorder (excluding childhood febrile convulsions) or epilepsy.
* Active liver disease.
* Any contraindication to the use of MC.
* Inflammatory Bowel Disease (IBD).

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
correlation of microbiome composition or serum metabolomics with pain reduction | Three Months
  Any correlation of the gut microbiome composition or serum metabolomics with pain reduction following a 3-months treatment period with cannabis oil.

SECONDARY OUTCOMES:
Pain Intensity | Three Months
  Change in pain intensity as measured by the Numeric Rating Scale
Change in sleep quality | Three Months
  Change in Pittsburgh Sleep Quality Index following 3 months of treatment with cannabis oil.
Change in quality of life | Three Months
  Change in Short-form health-questionnaire following 3 months of treatment with cannabis oil.
Change in anxiety and depression | Three Months
  Change in Hospital anxiety and depression scale following 3 months of treatment with cannabis oil.
Patient global impression of changes | Three Months
  Patient global impression of change following 3 months of treatment with cannabis oil.
Changes in gut microbiome and blood metabolites following 3 months treatment with cannabis oil | Three Months
  Changes in gut microbiome and blood metabolites following 3 months of treatment with cannabis oil will be measured using 16rRNA sequencing of stool and mass spectrometry of plasma.
correlation of microbiome composition and serum metabolomics with clinical measures | Three Months
  Significant correlations (using Kendall rank) of the relative abundance of measured gut bacteria and plasma metabolites with clinical measures including sleep, quality of life, anxiety, depression, and impression of change following a 3-month treatment period with cannabis oil.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Minerbi, MD-PhD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, raw data and analyses will be made available once the data analysis is complete and the study results are ready for peer review.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Estimated May 2027 for unlimited time.
Access Criteria: All non identified data will be made publicly available.